CLINICAL TRIAL: NCT00134472
Title: Therapeutic Strategy for Severe Head Trauma Patients With Mild Hypothermia and Estimation of Medical Expenses in Japan
Brief Title: Therapeutic Hypothermia for Severe Traumatic Brain Injury in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yamaguchi University Hospital (Other)
Collaborators: University Hospital Medical Information Network (Other); Japan Clinical Research Support Unit(J-CRSU) (Unknown)
Responsible Party: Principal Investigator, Tsuyoshi Maekawa, Honorary Professor, Yamaguchi University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H14-HEART-005; H15-HEART-01; H16-HEART-01
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Brain Injuries, Traumatic
Keywords: Hypothermia, induced; Traumatic Brain injuries; Anesthesia; Neuro-intensive care; neurochemistry
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypothermia

INTERVENTIONS:
Procedure: Therapeutic mild hypothermia — Keeping 32 - 34 degree celsius of core temperature at least for 72 hours.

SUMMARY:
The purpose of this trial is to determine if mild hypothermia therapy, for severe head trauma patients, improves neurological outcome.

DETAILED DESCRIPTION:
Mild hypothermia therapy shows protective effects for damaged brains of animals and post cardiac arrest patients. However, Clifton et al. reported that mild hypothermia has no protective effect for severe head trauma but has a risk of complications. In this study, all the participants must be treated with continuous monitoring of cardiac output and jugular venous oxygen saturation to get optimal physiological conditions. Adequate anesthesia such as neuroleptanesthesia is essential to maintain organ function and tissue microcirculation. Participants are randomly assigned to two groups of mild hypothermia (32.0 - 34.0 degree Celsius) and anti-hyperthermia (35.5 - 37.0 C). The body temperature must be kept for at least 72 hours. Hypothermia must be induced within 6 hours after traumatic brain injury. Glasgow outcome score at 6 months after injury and the total medical expenses of the two groups will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury; Glasgow coma score 4-8 (motor 1-5).
* Hypothermia or anti-hyperthermia must be induced within 6 hours after injury.

Exclusion Criteria:

* Systolic blood pressure < 90mmHg (after resuscitation)
* Thrombocytopenia (platelets [Plt] < 50,000/mm3)
* Pregnancy
* Preexisting medical conditions of severe hepatic dysfunction, heart failure or any other severe organ failure
* Deep drunkenness

Ages: 15 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2002-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Neurological outcome | six months after the onset
  Glasgow outcome score and neuropsychological performance at 6 months after injury.
Total medical expenses | whole duration of treatment
  Total medical expenses would be compared.

SECONDARY OUTCOMES:
Physiological data | each day during the treatment
Laboratory data | each day during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tsuyoshi Maekawa, MD, PhD, Principal Investigator — Yamaguchi University Hospital
Locations (43):
- Japan (43):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Chiba University Hospital, Chiba, Chiba
  - Chiba Emergency Medical Center, Chiba, Chiba
  - Ehime University Hospital, Tōon, Ehime
  - Ohta Nishinouchi Hospital, kooriyama, Fukushima
  - Gifu University Hospital, Gifu, Gifu
  - Sapporo Medical University, Sapporo, Hokkaido
  - The Hospital of Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Kanazawa University, Kanazawa, Ishikawa-ken
  - Iwate Medical University, Morioka, Iwate
  - Kagawa University Hospital, Kida, Kagawa-ken
  - St. Marianna University, School of Medicine, Kawasaki, Kanagawa
  - Kitasato University, Sagamihara, Kanagawa
  - Yokohama City Seibu Hospital, Yokohama, Kanagawa
  - Aizawa Hospital, Matsumoto, Nagano
  - Shinshu University Hospital, Matsumoto, Nagano
  - Nara Medical University, Kashihara, Nara
  - Oita University Faculty of Medicine, Ōita, Oita Prefecture
  - Kawasaki Medical University, Kurashiki, Okayama-ken
  - National Hospital Organization Osaka National Hospital, Cyuo, Osaka
  - Kansai Medical University, Moriguchi, Osaka
  - Osaka Mishima Emergency Medical Center, Takatsuki, Osaka
  - Saga Prefectural Hospital Kouseikan, Saga, Saga-ken
  - Saitama Medical Center, Kawagoe, Saitama
  - Shiga University of Medical Science, Ōtsu, Shiga
  - Saiseikai Utsunomiya Hospital, Utsunomiya, Tochigi
  - Tokushima University Hospital, Kuramoto, Tokushima
  - Nippon Medical School, Bunkyo, Tokyo
  - The University of Tokyo Hospital, Bunkyo, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Hachiōji, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro City, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Musashino Red Cross Hospital, Musashino, Tokyo
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
  - Showa University Hospital, Shinagawa, Tokyo
  - Tokyo Medical University, Shinjuku, Tokyo
  - Teikyo University Hospital, tabashi City, Tokyo
  - Nihon University Itabashi Hospital, tabashi City, Tokyo
  - Tama Nagayama Hospital, Nippon Medical School, Tama, Tokyo
  - Yamagata University Hospital, Yamagata, Yamagata
  - Advanced Medical Emergency and Critical Care Center, Yamaguchi University Hospital, Ube, Yamaguchi